CLINICAL TRIAL: NCT03808038
Title: Symptoms of Lower Urinary Tract Dysfunction Research Network (LURN) Protocol 2/Recall Study
Brief Title: Symptoms of Lower Urinary Tract Dysfunction Protocol 2/Recall Study
Status: Completed | Type: Observational
Sponsor: Arbor Research Collaborative for Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Michigan (Other); Northwestern University (Other); Duke University (Other); University of Iowa (Other); University of Washington (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: LURN Recall Study; U01DK097780 (NIH); U01DK097772 (NIH); U01DK097779 (NIH); U01DK099932 (NIH); U01DK100011 (NIH); U01DK100017 (NIH); U01DK097776 (NIH); U01DK099879 (NIH)
Record Dates: First submitted 2019-01-14; First posted 2019-01-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Lower Urinary Tract Symptoms; Bladder Symptoms; Recall; Lower Urinary Tract Dysfunction
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No Diary Group: Group completed daily questionnaires for four weeks, a weekly questionnaire at the end of each week, and a monthly questionnaire at the end of the study
  Interventions: Other: None- Observational Study
- Diary Start Group: Group completed bladder diaries in week 1, daily questionnaires in week 1, a weekly questionnaire at the end of each week, and a monthly questionnaire at the end of the study
  Interventions: Other: None- Observational Study
- Daily Start Group: Group completed daily questionnaires in week 1, bladder diaries in week 2, a weekly questionnaire at the end of each week, and a monthly questionnaire at the end of the study
  Interventions: Other: None- Observational Study

INTERVENTIONS:
Other: None- Observational Study — None- Observational Study

SUMMARY:
The purpose of this study is to advance the understanding of people who experience urinary and bladder problems. The investigators are interested in learning about people's experiences with urinary symptoms and how these symptoms will be managed. The investigators want to understand the important differences among people and what factors affect urinary and bladder problems. After all of the information is collected, the investigators will have a better understanding of how to improve the care and treatment for people who have urinary and bladder problems.

DETAILED DESCRIPTION:
This protocol is part of an overall effort to create a state-of-the-art resource for measuring patient-reported health for patients with lower urinary tract dysfunction (LUTD). The primary purpose of this resource, known as the LURN PRO Battery, is to comprehensively characterize the self-reported experiences of patients with LUTD for the purpose of enhancing efforts to characterize and explain important subtypes of patients with LUTD (phenotypes). Secondary purposes of the LURN PRO Battery, for which additional development work will be required, include developing better patient-reported endpoints for clinical trials, monitoring symptoms in the course of clinical care, and screening patients into important subgroups for purposes of tailored interventions.

Incorporating methods the investigators have used successfully in prior measure validation work, the investigators propose to conduct a diary study in which patients record their symptoms at various time points - at the end of each day, or across multiple days. The investigators also ask them to complete self-report measures with different recall periods (i.e., 3-day, 7-day, and 30-day recall), and will determine how well each of these correspond to daily experiences recorded in more frequent assessments (i.e., end-of-day and 3-day patient bladder diaries). These data will help LURN investigators to determine the most appropriate reporting period for specific symptoms. This study can also help to identify causes of differences that exist between shorter and longer recall periods.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 or older,
2. willing and able to give informed consent,
3. able to speak, read, and understand English,
4. able to reliably complete self-reported questionnaires online at specified times (i.e., may exclude those who do not keep a regular schedule of sleeping during night hours), and
5. experienced at least moderate severity and bother from at least 1 of the 7 targeted symptoms in the past 2 weeks and in the past 3 months

Exclusion Criteria:

1. dementia or other cognitive impairment that would interfere with study participation,
2. known pregnancy or delivery within past 6 months (women only)
3. planned change in medications to treat LUTS in the middle of the study time frame,
4. receiving active treatment for any malignancy (including maintenance medications),
5. received surgery with general or spinal/epidural anesthesia in the past 3 months or planned surgery during the study time frame
6. lower urinary tract instrumentation (e.g. self-catheterization or cystoscopy) in past 3 months or planned during the study time frame and
7. prostate biopsy in the past 3 months or planned during the study time frame

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with LUTS presenting to LURN clinical sites will be screened for participation based on the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Determine ideal recall period for LUTS symptoms | Through study completion - 30 days
  The investigators will administer and analyze the correspondence between patient's average daily recall of their LUTS utilizing seven, daily questionnaires, their weekly recall of self-reported LUTS using a 7-day recall questionnaire, as well as a questionnaire assessing their monthly LUTS recall in order to determine the best recall period to utilize when administering LUTS questionnaires in clinical settings.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P. Weinfurt, PhD, Study Chair — Duke University; Claire C. Yang, MD, Study Chair — University of Washington; Robert M. Merion, MD, FACS, Principal Investigator — Arbor Research Collaborative for Health - DCC
Locations (6):
- United States (6):
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
We do not plan to make IPD available.